CLINICAL TRIAL: NCT01205490
Title: Changes in Cerebral Blood Flow With Spinal Manipulative Therapy vs. Voluntary Motion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Canadian Memorial Chiropractic College (Other)
Collaborators: Canadian Medical Protective Association (Other); NCMIC (Unknown)
Responsible Party: Greg Wells, University of Toronto
Masking: Single | Purpose: Basic Science
Other Study IDs: 102026
Record Dates: First submitted 2010-09-17; First posted 2010-09-20 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Vertebral Artery Dissection; Cerebrovascular Accident; Cerebrovascular Stroke
MeSH Terms: conditions — Vertebral Artery Dissection; Stroke | interventions — Manipulation, Spinal

STUDY DESIGN:
Who Masked: Outcomes Assessor

INTERVENTIONS:
Other: head positions and spinal manipulation — Each subject will then undergo a baseline MRI in a head neutral position (0 degrees rotation). They will then be placed in head rotation (45 degrees) to the non-dominant and undergo a MRI. Maximum rotation to the side with MRI will follow. Finally, each subject will receive an upper cervical rotary manipulation to the non-dominant side with MRI immediately after. A total of 4 test conditions will be evaluated (rest, 45 degree, maximal, post-manipulation). The manipulation will be performed by an experience practitioner on a bed just outside the MRI room in supine position. A controlled impulse load will be applied and the head/neck returned to neutral position. Prior to each maneuver, the subject will be queried on their comfort, condition and willingness to continue

SUMMARY:
The investigators are performing a study to determine whether changes in blood flow occur in the neck and back of the brain following a series of head positions and a manipulation of the upper neck. Each participant will be asked to undergo a series of MRI's to evaluate whether there are any changes in blood flow resulting from any of the head positions or manipulation. The study will be conducted over a period of 1 day and each participant can anticipate the testing to take approximately 120 minutes.

DETAILED DESCRIPTION:
The goal is to further investigate the cerebrovascular hemodynamic consequences of cervical spine positions, including rotation and manipulation in-vivo under clinically relevant circumstances using two advanced forms of MRI technology on the VA and posterior cerebral vessels. According to the knowledge of the investigators, a study utilizing MRI and functional blood oxygen level dependent (fBOLD) imaging to examine blood flow and perfusion, turbulence and evidence of micro-trauma within these vessels has yet to be conducted.

ELIGIBILITY:
Inclusion/Exclusion Criteria

1. Enrolled and matriculated as a student in the Canadian Memorial Chiropractic College.
2. Healthy asymptomatic male patients who would otherwise receive cervical manipulation on a regular basis as a part of their normal learning experience and will have had a cervical manipulation in the last 3 months.
3. Sufficient English language ability to complete study questionnaires (see appendix).
4. No history of disabling neck, arm or headache pain within the last 6 months.
5. No current or prior history of neurological symptoms including, facial or extremity weakness, abnormal sensation to the face, body or extremities, uncontrolled movements, abnormal gait, dizziness, unexplained nausea/vomiting, difficulty with speaking or swallowing.
6. Subjects will have had no prior history of head trauma or prior history of surgery to the neck region.
7. No history of claustrophobia, metallic implants or tattoos to ensure compatibility with MRI requirements.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
change in advanced magnetic resonance imaging | immediately after head positions.
  A change in vertebral, posterior cerebellar and collateral arterial blood flow associated with various head positions and an upper cervical manipulation will be measured using blood oxygen level dependent (BOLD). A BOLD MRI generates a signal by tracking changes in the local oxyhemoglobin to deoxyhemoglobin ratio. Signal changes are due to a combination of altered microvascular perfusion, blood volume, and fluctuations in cellular metabolism. It will also provide more sensitivity in determining the impact of changes in blood flow during the various head positions.

CONTACTS AND LOCATIONS:
Overall Officials: Greg Wells, PhD, Principal Investigator — University of Toronto; Jairus Quesnele, BSc, DC, Principal Investigator — Canadian Memorial Chiropractic College; John J Triano, DC, PhD, Study Chair — Canadian Memorial Chiropractic College; Michael Noseworthy, PhD, Study Director — McMaster University
Locations (1):
- St. Joseph Healthcare, Research Imaging Institute, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Boyle E, Cote P, Grier AR, Cassidy JD. Examining vertebrobasilar artery stroke in two Canadian provinces. J Manipulative Physiol Ther. 2009 Feb;32(2 Suppl):S194-200. doi: 10.1016/j.jmpt.2008.11.019. PMID 19251064
- [Background] Cassidy JD, Boyle E, Cote P, He Y, Hogg-Johnson S, Silver FL, Bondy SJ. Risk of vertebrobasilar stroke and chiropractic care: results of a population-based case-control and case-crossover study. J Manipulative Physiol Ther. 2009 Feb;32(2 Suppl):S201-8. doi: 10.1016/j.jmpt.2008.11.020. PMID 19251066
- [Background] Rubinstein SM, Peerdeman SM, van Tulder MW, Riphagen I, Haldeman S. A systematic review of the risk factors for cervical artery dissection. Stroke. 2005 Jul;36(7):1575-80. doi: 10.1161/01.STR.0000169919.73219.30. Epub 2005 Jun 2. PMID 15933263
- [Background] Zaina C, Grant R, Johnson C, Dansie B, Taylor J, Spyropolous P. The effect of cervical rotation on blood flow in the contralateral vertebral artery. Man Ther. 2003 May;8(2):103-9. doi: 10.1016/s1356-689x(02)00155-8. PMID 12890438
- [Background] Cagnie B, Jacobs F, Barbaix E, Vinck E, Dierckx R, Cambier D. Changes in cerebellar blood flow after manipulation of the cervical spine using Technetium 99m-ethyl cysteinate dimer. J Manipulative Physiol Ther. 2005 Feb;28(2):103-7. doi: 10.1016/j.jmpt.2005.01.005. PMID 15800509
- [Background] Mitchell JA. Changes in vertebral artery blood flow following normal rotation of the cervical spine. J Manipulative Physiol Ther. 2003 Jul-Aug;26(6):347-51. doi: 10.1016/S0161-4754(03)00074-5. PMID 12902962
- [Background] Johnson C, Grant R, Dansie B, Taylor J, Spyropolous P. Measurement of blood flow in the vertebral artery using colour duplex Doppler ultrasound: establishment of the reliability of selected parameters. Man Ther. 2000 Feb;5(1):21-9. doi: 10.1054/math.1999.0227. PMID 10688956
- [Background] Sakaguchi M, Kitagawa K, Hougaku H, Hashimoto H, Nagai Y, Yamagami H, Ohtsuki T, Oku N, Hashikawa K, Matsushita K, Matsumoto M, Hori M. Mechanical compression of the extracranial vertebral artery during neck rotation. Neurology. 2003 Sep 23;61(6):845-7. doi: 10.1212/01.wnl.0000078081.12097.ae. PMID 14504337
- [Background] Haynes MJ. Doppler studies comparing the effects of cervical rotation and lateral flexion on vertebral artery blood flow. J Manipulative Physiol Ther. 1996 Jul-Aug;19(6):378-84. PMID 8864968
- [Background] Licht PB, Christensen HW, Hojgaard P, Hoilund-Carlsen PF. Triplex ultrasound of vertebral artery flow during cervical rotation. J Manipulative Physiol Ther. 1998 Jan;21(1):27-31. PMID 9467098
- [Background] Licht PB, Christensen HW, Svendensen P, Hoilund-Carlsen PF. Vertebral artery flow and cervical manipulation: an experimental study. J Manipulative Physiol Ther. 1999 Sep;22(7):431-5. doi: 10.1016/s0161-4754(99)70030-8. PMID 10519558
- [Background] Bendick PJ, Jackson VP. Evaluation of the vertebral arteries with duplex sonography. J Vasc Surg. 1986 Mar;3(3):523-30. doi: 10.1067/mva.1986.avs0030523. PMID 3512861